CLINICAL TRIAL: NCT01646047
Title: Effects of a Novel Dietary Supplement on Visual Function in Patients With Diabetes With and Without Early Diabetic Retinopathy
Brief Title: Diabetes Visual Function Supplement Study
Acronym: DiVFuSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZeaVision, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20112190
Record Dates: First submitted 2012-07-03; First posted 2012-07-20 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus - Type 1; Diabetes Mellitus - Type 2; Non-proliferative Diabetic Retinopathy
Keywords: diabetes; diabetic retinopathy; nutritional supplements; visual function; macular pigment; macular threshold sensitivity; contrast sensitivity; color vision; optical coherence tomography
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- supplement - no retinopathy (Experimental): subjects receiving active supplement and with no retinopathy based on clinical examination
  Interventions: Dietary Supplement: multi-component nutritional supplement capsules
- placebo - no retinopathy (Placebo Comparator): patients receiving placebo and who have no diabetic retinopathy based on clinical examination
  Interventions: Dietary Supplement: multi-component dietary supplement
- supplement - retinopathy (Experimental): patients receiving the active supplement and who have mild to moderate non-proliferative diabetic retinopathy based on clinical examination
  Interventions: Dietary Supplement: multi-component nutritional supplement capsules
- placebo - retinopathy (Placebo Comparator): patients receiving placebo and who have mild to moderate non-proliferative diabetic retinopathy based on clinical examination
  Interventions: Dietary Supplement: multi-component dietary supplement

INTERVENTIONS:
Dietary Supplement: multi-component nutritional supplement capsules — two capsules containing nutritional supplements per day for 6 months (vitamin C, mixed tocopherols/tocotrienols, vitamin D, fish oil, lutein, zeaxanthin, pine bark extract, benfotiamine, green tea extract, curcumin)
  Arms: supplement - no retinopathy; supplement - retinopathy
Dietary Supplement: multi-component dietary supplement — placebo capsules
  Other Names: two placebo capsules per day for six months
  Arms: placebo - no retinopathy; placebo - retinopathy

SUMMARY:
This study will evaluate the effects of a novel multi-component dietary supplement on the visual function and retinal structure of patients with diabetes with both no diabetic retinopathy and mild to moderate diabetic retinopathy. This is a placebo-controlled trial and neither subjects nor examiners will know if any given subject is taking active supplement or placebo.

The hypothesis is that the supplement will improve visual function and retinal structure in subjects on active supplement

DETAILED DESCRIPTION:
Adult patients with either type 1 or type 2 diabetes will be enrolled with baseline measurement of visual acuity, contrast sensitivity, color vision, threshold macular perimetry, macular pigment optical density, optical coherence tomography, glycosylated hemoglobin, blood lipids and serum vitamin D status. A multi-component dietary supplement containing ingredients currently available over the counter in the US will be taken for six months and repeat measurements of the above parameters obtained.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus diagnosed at least 5 years
* age greater than or equal to 18 years
* English speaker

Exclusion Criteria:

* proliferative diabetic retinopathy or severe non-proliferative retinopathy
* clinically significant macular edema
* corrected visual acuity less than 20/30 in either eye
* diagnosis of other serious eye disease (glaucoma, age-related maculopathy)
* less than 18 years old
* non-English speaker
* no known allergy or sensitivity to any supplement ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Changes in visual function | At baseline and again at six months
  Change in contrast sensitivity, color vision and macular perimetry thresholds

SECONDARY OUTCOMES:
Changes in serum markers | At baseline and again at six months
  Changes in glycosylated hemoglobin, serum lipids, serum vitamin D (all subjects) and the serum inflammatory cytokine, tumor necrosis factor-alpha (subjects with retinopathy)
Changes in retinal structure | At baseline and again at 6 months
  Changes in optical coherence tomography and macular pigment optical density

CONTACTS AND LOCATIONS:
Overall Officials: Alan P. Chous, O.D., Principal Investigator — Chous Eye Care Associates
Locations (1):
- Chous Eye Care Associates, Tacoma, Washington, United States

REFERENCES:
- [Derived] Robertson NU, Schoonees A, Brand A, Visser J. Pine bark (Pinus spp.) extract for treating chronic disorders. Cochrane Database Syst Rev. 2020 Sep 29;9(9):CD008294. doi: 10.1002/14651858.CD008294.pub5. PMID 32990945
- [Derived] Chous AP, Richer SP, Gerson JD, Kowluru RA. The Diabetes Visual Function Supplement Study (DiVFuSS). Br J Ophthalmol. 2016 Feb;100(2):227-34. doi: 10.1136/bjophthalmol-2014-306534. Epub 2015 Jun 18. PMID 26089210